CLINICAL TRIAL: NCT06864559
Title: Comparison of Three Types of Sutures in Oral Surgery. Study of Bacterial Colonization, Tissue Reaction and Clinical Characteristics: Randomized Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jose Manuel Alarcón Cordovilla, DDS (University of Granada), MSc (Oral Surgery), Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2028/CEIH/2021
Record Dates: First submitted 2025-02-22; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Wound Healing Complication; Oral Surgery; Third Molar Extraction; Oral Infection
MeSH Terms: interventions — Surgery, Oral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Suture 1: Silk. (Other): Silk suture.
  Interventions: Other: To Compare 3 different suture materials used in oral surgery
- Suture 2: Non-absorbable polyamide monofilament. (Other): Non-absorbable polyamide monofilament.
  Interventions: Other: To Compare 3 different suture materials used in oral surgery
- Suture 3: Non-resorbable expanded polytetrafluoroethylene. (Other): Non-resorbable expanded polytetrafluoroethylene.
  Interventions: Other: To Compare 3 different suture materials used in oral surgery

INTERVENTIONS:
Other: To Compare 3 different suture materials used in oral surgery — To compare bacterial colonization, tissue reaction and clinical characteristics such as wound healing and patient postoperative outcomes in 3 different suture materials used in oral surgery.
  Other Names: 2028/CEIH/2021

SUMMARY:
Considering the wide variety of surgical sutures currently marketed in the field of Dentistry, it was decided to conduct a study comparing the microbial adhesion and antibacterial activity of three different types of sutures used in Oral Surgery (Silk, non-absorbable polyamide monofilament and non-absorbable expanded polytetrafluoroethylene).

DETAILED DESCRIPTION:
The general or primary objective is:

• To compare 3 non-absorbable suture materials used in oral surgery: silk, polyamide monofilament and expanded polytetrafluoroethylene.

The specific or secondary objectives are:

* To evaluate how each type of suture influences wound healing and the patient's postoperative period.
* To study bacterial colonization in each type of suture.
* To determine the tissue reaction and clinical characteristics of each suture.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for extraction of a third lower molar retained in an unfavorable position that requires a bayonet incision in the surgical procedure.
* Age: patients aged 18 years or older.
* ASA I patients (Classification of the American Society of Anesthesiology, 1979): healthy patients who tolerate stress well, without systemic pathology, no anxiety and in whom a therapeutic modification is not necessary.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Smoking patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Bacterial colonization | 7 days.
  Microbiological analysis: CFU and qPCR bacterial count.
Level of inflammation | 7 days.
  The degree of soft tissue inflammation was assessed using Visual Analogue Scale (VAS).